CLINICAL TRIAL: NCT01978327
Title: Single-blind, Randomised, Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Repeat Doses of GSK2647544 and Its Potential Pharmacokinetic Interaction With Simvastatin in Healthy Volunteers
Brief Title: GSK2647544 RD, DDI in Healthy Young and Elderly Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Given the strength of CYP3A4 inhibition observed in Cohort 1, there is no rationale to investigate higher doses of GSK2647544 in the following two cohorts
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 200592
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; GSK2647544; drug-drug interaction; healthy subjects; Lp-PLA2; simvastatin
MeSH Terms: conditions — Alzheimer Disease | interventions — GSK2647544; Drug Interactions

STUDY DESIGN:
Who Masked: Participant

ARMS (4):
- GSK2647544 (Experimental): The planned repeat doses of GSK2647544 are 80 mg bid, 200 mg bid, and 350 mg bid
  Interventions: Drug: GSK2647544
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: GSK2647544
- simvastatin (Experimental): for drug-drug interaction
  Interventions: Drug: drug-drug interaction
- simvastatin co-dosed with GSK2647544 (Experimental): for drug-drug interaction
  Interventions: Drug: drug-drug interaction

INTERVENTIONS:
Drug: GSK2647544 — repeat dose
  Arms: GSK2647544; Placebo
Drug: drug-drug interaction — drug-drug interaction
  Arms: simvastatin; simvastatin co-dosed with GSK2647544

SUMMARY:
GSK2647544 is an orally available, selective inhibitor of Lp PLA2 that is being developed for the treatment of Alzheimer's disease. The current study is a single-blind, randomised, placebo-controlled, 4-cohort study to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of repeat doses of GSK2647544. Cohorts 1, 2 and 3 will evaluate escalating doses of GSK2647544 in young healthy volunteers for 7 days, 7 days, and 14 days, respectively. Cohort 4 will evaluate repeat doses of GSK2647544 in healthy elderly volunteers for 14 days. Additionally, Cohorts 1 and 3 will include an assessment of potential drug-drug interaction with simvastatin to examine CYP3A4 inhibition by GSK2647544.

ELIGIBILITY:
Inclusion Criteria:

* Males and females who are 18 to 64 years of age inclusive, defined as young subjects in this study, are eligible for Cohorts 1-3 only
* Males and females who are ≥65 years of age, defined as elderly subjects in this study, are eligible for Cohort 4 only
* Healthy as determined by a responsible and experienced physician
* A female subject is eligible to participate if she is of non-childbearing potential
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods
* Body weight > 50 kg (110 pounds) and body mass index (BMI) between 19 and 32
* Aspartate aminotransferase (AST), Alanine transaminase (ALT), alkaline phosphatase and bilirubin <= 1.5xUpper Limit of Normal (ULN)
* Average of triplicate QTcB values and average of triplicate QTcF values must both < 450 msec
* Capable of giving written informed consent

Exclusion Criteria:

* Subjects with Lp-PLA2 activity <=20 nanomole/minute/milliliter (mL)(for subjects with 2 known birth parents of at least 50% Japanese, Chinese, or Korean ancestry)
* History of asthma, anaphylaxis or anaphalactoid reactions, severe allergic responses
* History of hypercoagulable state or history of thrombosis
* History of biliary tract disease including a history of liver disease with elevated liver function tests of known or unknown etiology
* Positive Human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C at screening
* History of regular use of tobacco or nicotine-containing products within 6 months of the study
* Unable to abstain from alcohol or caffeine or xanthine-containing products for 24 h prior to the start of dosing
* Unable to refrain from use of prescription or non-prescription drugs and vitamins within 7 days or 5 half-lives (whichever is longer) prior to administration of study
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening (Note: This applies to healthy young subjects screened for Cohorts 1-3 only. Healthy elderly subjects for cohort 4 who are social smokers must give up smoking for the period that they will be on the unit)
* positive pre-study drug/alcohol screen
* Unable to refrain from consumption of Seville oranges, grapefruit or grapefruit juice within 7 days prior to the first dose of study medication until the follow-up visit
* Subjects who have taken statins, medicines that are contraindications of statins, know potent inhibitiors or inducers of CYP3A4 in the 4 weeks or 5 half-lives (whichever is longer) prior to screening and are not able to discontinue use throughout participation in the clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-11-22 (Actual); Primary Completion 2014-03-03 (Actual); Study Completion 2014-03-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of GSK2647544 as assessed by number of subjects with adverse events (AE)s | up to 19 days in each dosing session
  Safety and tolerability parameters will include recording of AEs
Safety and tolerability of GSK2647544 as assessed by change from Baseline in laboratory values | up to 15 days in each dosing session
  Safety and tolerability parameters will include laboratory (haematology, clinical chemistry, urinalysis) values at Screening, Day-1, Day 1 to up to Day 15 and Follow-up (7-14 days post-last dose)
Safety and tolerability of GSK2647544 as assessed by change from Baseline in ECG readings | up to 19 days in each dosing session
  Safety and tolerability parameter will include the electrocardiogram (ECG) readings at Screening, Day -1, Day 1 to up to Day 19, and follow-up (7-14 days post-last dose)
Safety and tolerability of GSK2647544 as assessed by change from Baseline in Telemetry ECG parameters | 2 days in Cohorts 1, 2 and 4; 3 days in Cohort 4
  Safety and tolerability parameter will include the Telemetry ECG readings from 30 minutes pre-dosing till 24 hours post-dosing
Safety and tolerability of GSK2647544 as assessed by change from Baseline in vital signs | up to 19 days in each dosing session
  Vital signs measurement include systolic and diastolic blood pressure and pulse rate at Screening, Day -1, Day 1 to up to Day 19, and Follow-up (7-14 days post-last dose)
Safety and tolerability of GSK2647544 as assessed by Columbia Suicide Severity Rating Scale (C-SSRS) | 4 days in Cohorts 1 and 2; 8 days in Cohorts 3 and 4
  C-SSRS will be measured at Screening, Day-1, dispersed days during dosing sessions, prior to discharge, and Follow-up (7-14 days post-last dose)
Peak plasma concentration (Cmax) of GSK2647544 | up to 17 days in GSK2647544 dosing sessions
  To assess PK profile of GSK2647544, Cmax of GSK2647544 will be measured
Time of peak plasma concentration (tmax) of GSK2647544 | up to 17 days in GSK2647544 dosing sessions
  To assess PK profile of GSK2647544, tmax of GSK2647544 will be measured
Area under the time concentration curve (AUC) of GSK2647544 | up to 17 days in GSK2647544 dosing sessions
  To assess PK profile of GSK2647544, AUC of GSK2647544 will be measured
Terminal half-life (t½ ) of GSK2647544 | up to 17 days in GSK2647544 dosing sessions
  To assess PK profile of GSK2647544, t1/2 of GSK2647544 will be measured
Time of peak plasma concentration (tmax) of simvastatin | 4 days in Cohorts 1 and 3
  To assess the effect of GSK2647544 on PK profile of simvastatin, tmax of simvastatin will be measured
Area under the time concentration curve (AUC) of simvastatin | 4 days in Cohorts 1 and 3
  To assess the effect of GSK2647544 on PK profile of simvastatin, AUC of simvastatin will be measured

SECONDARY OUTCOMES:
Predose plasma lipoprotein-associated phospholipase A2 (Lp-PLA2) activity and postdose Lp-PLA2 activity | up to 18 days in GSK2647544 dosing sessions
  Lp-PLA2 activity will be measured at Days 1, 2, 3 and 4 in GSK2647544 single dose sessions; it will be measured at Days 1, 3, 4, 5, 7, 10, 14, 15, 16, 17 and 18 in GSK2647544 repeat dose sessions

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Harrow, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 200592 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/200592?search=study&study_ids=200592#rs
- Available data/document: Dataset Specification: 200592 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 200592 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 200592 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 200592 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 200592 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 200592 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 200592 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register